CLINICAL TRIAL: NCT05141929
Title: Effect of Web-Based Education Related to Gestational Diabetes Mellitus on Women Health Management Self Efficacy and Maternal-Fetal-Neonatal Results
Brief Title: Effect of Web-Based Education on Gestational Diabetes Mellitus and Health Management Self Efficacy
Acronym: GDM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Nuran Nur Aypar Akbağ, Director, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2908-GOA-2019/01-25
Record Dates: First submitted 2021-10-25; First posted 2021-12-02 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Pregnancy Complications; Efficacy, Self
Keywords: Gestational Diabetes Mellitus; self efficacy; web based education
MeSH Terms: conditions — Pregnancy Complications; Diabetes, Gestational

STUDY DESIGN:
Intervention Model Description: A randomized control study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): web based education and routine clinical procedure
  Interventions: Behavioral: web based education
- control group (No Intervention): only routine clinical procedure

INTERVENTIONS:
Behavioral: web based education — In addition to routine care, web-based education was offered to pregnant women with Gestational Diabetes Mellitus.
  Other Names: only routine clinical procedure
  Arms: intervention group

SUMMARY:
This randomized controlled study aimed to examine the effect of web-based education related to Gestational Diabetes Mellitus on women health management self-efficacy and maternal-fetal-neonatal results.

DETAILED DESCRIPTION:
Objective: To examine the effect of web-based education related to Gestational Diabetes Mellitus on women health management self-efficacy and maternal-fetal-neonatal results.

Design: Randomized controlled study. Patients: Thirty one pregnant women were included in the intervention group and thirty four pregnant women in the control group.

Interventions: For 8 weeks, web-based education for Gestational Diabetes Mellitus was offered to pregnant women who diagnosed with Gestational Diabetes Mellitus for the first time. The data were collected before web-based education, after web-based education and postpartum between 4-12 weeks at three different times. Control group was offered routine clinical procedure.

Main Outcome Measures: health management self efficacy (primary outcomes), maternal-fetal-neonatal results (secondary outcome).

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older
* Being primigravida or multigravida
* Getting a diagnosis of Gestational Diabetes Mellitus
* Having a gestational week between 24-28
* Having a single fetus
* Ability to use the Internet (Computer, tablet, smart phone, etc.)
* Voluntary participation in the research

Exclusion Criteria:

* Having a diagnosis of Type 1 and Type 2 Diabetes Mellitus
* Having another chronic disease
* Having a visual or hearing impairment
* Having a psychiatric medical diagnosis
* Having a diagnosis of risky pregnancy not related to GDM

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Change from Self Rated Abilities for Health Practices levels in pregnant women with GDM | Change in Self Rated Abilities for Health Practices levels up to postpartum 12th week
  Self Rated Abilities for Health Practices Scale: Self Rated Abilities for Health Practices Scale: The 5-point Likert scale was adapted for Turkish version by Aypar Akbağ and Aluş Tokat (Aypar Akbağ and Aluş Tokat, 2021). The scale consists of 4 sub-dimensions: "Exercise"," Responsible Health Practices", "Psychological Well Being" and "Nutrition". (from 0 (not at all) to 4 (completely). The scale total-score ranged between 0 and 112, while subscale total-scores ranging from 0 to 28 points. The higher scores from the scale indicate higher self-efficacy levels for the health applications.

SECONDARY OUTCOMES:
Rate of maternal-fetal-neonatal complications in pregnant women with GDM | Change in rate of maternal, fetal and neonatal complications up to postpartum 12th week
  The chart was used to evaluate the maternal (ketoacidosis, preeclampsia, polyhydramnios, preterm labor, vaginal or urinary infection), fetal (macrosomia, Intrauterine Growth Retardation) and neonatal (neonatal hypoglycemia, polycythemia and neonatal hyperbilirubinemia, duration of treatment for hyperbilirubinemia, Respiratory Distress Syndrome (RDS), hypothermia, dehydration) complications of Gestational Diabetes Mellitus. Complications during pregnancy and postpartum period were followed up. Complication follow-up was done by contacting the intervention group via the website. In the control group, complication follow-up was obtained by phone calls.

CONTACTS AND LOCATIONS:
Overall Officials: Nuran N Aypar Akbağ, Dr, Study Director — Karamanoğlu Mehmetbey University; Merlinda Aluş Tokat, Dr, Study Director — Dokuz Eylul University
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) is planned to be shared after the publication of the article.

REFERENCES:
- [Derived] Akbag NNA, Tokat MA. Effects of web-based gestational diabetes mellitus education on health management self-efficacy, treatment modality, and maternal-fetal-neonatal outcomes: A randomized controlled trial. Health Care Women Int. 2025 Dec 18:1-22. doi: 10.1080/07399332.2025.2597240. Online ahead of print. PMID 41412825